CLINICAL TRIAL: NCT05422469
Title: Neurobehavioral Investigations of Approach Dynamics in the Ventral Striatum
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Sameer Sheth, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 56119
Record Dates: First submitted 2022-05-27; First posted 2022-06-16 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Obsessive-Compulsive Disorder (OCD)
Keywords: Deep Brain Stimulation (DBS); Treatment Resistant OCD; Intractable OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Medtronic Percept RC neurostimulator (Experimental)
  Interventions: Device: Medtronic Percept RC neurostimulator

INTERVENTIONS:
Device: Medtronic Percept RC neurostimulator — Medtronic SenSight directional DBS leads and implanted pulse generators (IPGs) will be implanted

SUMMARY:
Traditional strategies for diagnosing psychiatric disorders focus on definitions based on constellations of co-occurring symptoms. Tracking symptom severity across therapy arcs relies on administering scales that again ask questions about symptoms. These strategies have allowed some degree of standardization but suffer from having a phenomenological rather than mechanistic foundation (in terms of diagnosis) as well as subjectivity and temporal sparseness (in terms of measurement).

The investigators apply a transdiagnostic framework based on the neurobiological concept of approach behavior. Several psychiatric disorders (including OCD, uni- and bipolar depression, PTSD and anxiety disorders, and addiction disorders) are characterized by dysfunction in approach behavior. The investigators study the neurobehavioral basis of approach dysfunction in a cohort of individuals with severe OCD and bipolar disorder (BD). To study these behaviors, the investigators deploy a suite of wearables and peripherals (Oura ring, Apple Watch, iPhone, audioband) that allow continuous and dense measurement of behaviors relevant to the approach hypothesis: socialization, activity, and sleep patterns. The investigators perform these measurements in two selected environments. One is a novel apartment-style setting (neurobehavioral unit, NBU) that combines the high-bandwidth data acquisition capability of a lab with the naturalistic relevance and comfort of the home. The second is the truly natural and maximally ethologically relevant setting of the ambulatory "home" environment in which people spend the majority of their time.

The participants will be individuals planned for deep brain stimulation (DBS) implant for their OCD or BD. The bi-directional (stimulate as well as record) nature of the DBS systems will allow neural recordings that the investigators will synchronize with the behavioral data streams. The investigators will apply predictive computational models in conjunction with the causal manipulation provided by stimulation to test mechanistic hypothesis relating neurophysiology, behavior, and clinical status. In Aim 1, The investigators study reward-driven decision making by employing an augmented reality approach-avoidance task in the NBU. In Aim 2, the investigators test the neurobehavioral models' ability to predict clinical status from passively (and therefore low burden to patient-participants) acquired data in the "home" environment. In Aim 3, the investigators identify neural predictors of the patterns of sleep dysregulation associated with these disorders using the unique environment of the NBU. In Aim 4, the investigators examine critical concepts of ethics and ethology that arise with this new field of naturalistic, chronic brain-behavior relationship investigation.

The investigators hope that methods validated and lessons learned in this project will improve understanding of the mechanistic basis of a range of psychiatric disorders and thereby allow greater rational design of therapeutic delivery.

DETAILED DESCRIPTION:
Traditional strategies for diagnosing psychiatric disorders focus on definitions based on constellations of co-occurring symptoms. Tracking symptom severity across therapy arcs relies on administering scales that again ask questions about symptoms. These strategies have allowed some degree of standardization but suffer from having a phenomenological rather than mechanistic foundation (in terms of diagnosis) as well as subjectivity and temporal sparseness (in terms of measurement).

The investigators apply a transdiagnostic framework based on the neurobiological concept of approach behavior. Several psychiatric disorders (including OCD, uni- and bipolar depression, PTSD and anxiety disorders, and addiction disorders) are characterized by dysfunction in approach behavior. The investigators study the neurobehavioral basis of approach dysfunction in a cohort of individuals with severe OCD and bipolar disorder (BD). To study these behaviors, the investigators deploy a suite of wearables and peripherals (Oura ring, Apple Watch, iPhone, audioband) that allow continuous and dense measurement of behaviors relevant to the approach hypothesis: socialization, activity, and sleep patterns. The investigators perform these measurements in two selected environments. One is a novel apartment-style setting (neurobehavioral unit, NBU) that combines the high-bandwidth data acquisition capability of a lab with the naturalistic relevance and comfort of the home. The second is the truly natural and maximally ethologically relevant setting of the ambulatory "home" environment in which people spend the majority of their time.

The participants will be individuals planned for deep brain stimulation (DBS) implant for their OCD or BD. The bi-directional (stimulate as well as record) nature of the DBS systems will allow neural recordings that the investigators will synchronize with the behavioral data streams. The investigators will apply predictive computational models in conjunction with the causal manipulation provided by stimulation to test mechanistic hypothesis relating neurophysiology, behavior, and clinical status. In Aim 1, The investigators study reward-driven decision making by employing an augmented reality approach-avoidance task in the NBU. In Aim 2, the investigators test the neurobehavioral models' ability to predict clinical status from passively (and therefore low burden to patient-participants) acquired data in the "home" environment. In Aim 3, the investigators identify neural predictors of the patterns of sleep dysregulation associated with these disorders using the unique environment of the NBU. In Aim 4, the investigators examine critical concepts of ethics and ethology that arise with this new field of naturalistic, chronic brain-behavior relationship investigation.

The investigators hope that methods validated and lessons learned in this project will improve understanding of the mechanistic basis of a range of psychiatric disorders and thereby allow greater rational design of therapeutic delivery.

ELIGIBILITY:
Inclusion Criteria:

* Planned for DBS for OCD (via clinical pathway, FDA HDE, IRB) or BD (via BRAIN-funded UH3 trial)
* Agrees to study activities in NBU and "home" environments

Exclusion Criteria:

- Planned to receive non-rechargeable DBS generator

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-08 (Estimated); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Change in Yale-Brown Obsessive-Compulsive Scale (YBOCS) Score | Through study completion, an average of 14 months
  Severity of depression symptoms. Changes in the Yale-Brown Obsessive Compulsive Scale survey/questionnaire. YBOCS is an assessment to rate symptoms of OCD on a scale of 0-50 (with a higher number indicating a more severe outcome ratings of OCD and 0 indicated no symptoms of OCD).
Change in Hamilton Depression Inventory (HAM-D) Score | Through study completion, an average of 14 months
  Severity of depression symptoms. Changes in the Hamilton Depression Inventory (HAM-D) score. HAM-D is an assessment to rate symptoms of depression on a scale of 0-52 (with a higher number indicating a more severe outcome ratings of depression and 0 indicated no symptoms of depression).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Brown University, Providence, Rhode Island
  - Baylor College of Medicine, Houston, Texas